CLINICAL TRIAL: NCT01821495
Title: A Randomized Controlled Study of Dendritic and Cytokine-induced Killer Cells (DC-CIK) Treatment in Patients With Staging Ⅱ-Ⅲ of Nasopharyngeal Carcinoma
Brief Title: Study of DC-CIK to Treat NPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Weiliang Sun, investigator, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPC-01
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: NPC,DC-CIK
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (No Intervention): After accepting concurrent radiotherapy and chemotherapy, patients will just regularly follow up.
- A (Experimental): After accepting concurrent radiotherapy and chemotherapy, patients will receive 3 cycles of Dendritic and Cytokine-induced Killer Cells (DC-CIK)treatment.
  Interventions: Biological: DC-CIK; Biological: Dendritic and Cytokine-induced Killer Cells

INTERVENTIONS:
Biological: DC-CIK
  Arms: A
Biological: Dendritic and Cytokine-induced Killer Cells — Concurrent of radiotherapy and chemotherapy plus 3 cycles of Dendritic and Cytokine-induced Killer Cells(DC-CIK) treatment
  Other Names: DC-CIK
  Arms: A

SUMMARY:
Concurrent of radiotherapy and chemotherapy is the main treatment method for patients with nasopharyngeal carcinoma (NPC). However, Relapse remains the major cause of treatment failure. A series of studies reported that dendritic and cytokine-induced killer cells (DC-CIK) have a broad anti-tumor spectrum. We suppose that DC-CIK will improve the prognosis of NPC. In this study, the patients with NPC will be treated with DC-CIK cells after concurrent of chemotherapy and radiotherapy. The purpose of this study is to evaluate the efficacy of DC-CIK for NPC.

DETAILED DESCRIPTION:
About 60 patients with staging Ⅱ-Ⅲ of NPC, after accepting concurrent radiotherapy and chemotherapy, will be randomly divided into group A (receive DC-CIK treatment) or group B (just regularly follow up), and the randomize ratio will be 1:1. Patients in group A will receive 2-3 cycles of DC-CIK cells treatment (every 4 weeks). Patients in group B will have no anti-tumor therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with staging Ⅱ-Ⅲ of NPC;
2. Patients who had completed concurrent of radiotherapy and chemotherapy;
3. Patients who have a life expectancy of at least 12 weeks;
4. Eastern Cooperative Oncology Group (ECOG) performance status was 0-1;
5. The bone marrow functioned normally (WBC > 4.0×109/L, Hb > 120 g/L, PLT > 100×109/L);
6. The ECG results were normal, and the liver and kidney were functional.

Exclusion Criteria:

1. Patients who had distant metastases by imaging studies;
2. Patients with uncontrolled infection; underlying disease that was severe or life-threatening;
3. Patients who were pregnant or lactating;
4. ECOG perform status ≥ 2;
5. Patients who are suffering from auto immune diseases or patients who need to accept glucocorticoid treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
progression-free survival(PFS) | 1 month

SECONDARY OUTCOMES:
overall survival(OS) | 1 month

OTHER OUTCOMES:
Laboratory findings | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Hanfeng Liu, Study Chair — Guangxi Medical University
Locations (1):
- Guangxi Medical University, Nanning, Guangxi, China